CLINICAL TRIAL: NCT02908516
Title: Safety and Efficacy of Oral Tranexamic Acid in Reducing Blood Loss and Transfusion in Femoral Neck, Intertrochanteric and Subtrochanteric Femur Fractures 100 FR 1 (2015-2)
Brief Title: Safety and Efficacy of Oral TXA in Reducing Blood Loss and Transfusion in Hip Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to inability to recruit and collect follow up outcome data.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2000020122
Record Dates: First submitted 2016-07-25; First posted 2016-09-21 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Hip Fractures; Blood Loss
MeSH Terms: conditions — Hip Fractures; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): Study subjects randomized to receive the TXA group will receive 3 oral capsules of 650 mg each of TXA for a total of 1.95 g. One dose will be given upon diagnosis of a hip fracture in the emergency department (ED) and a second dose will be given two hours prior to surgical incision.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Study subjects randomized to the placebo group will receive an equivalent dose of cellulose in 3 oral capsules. One dose will be given upon diagnosis of a hip fracture in the ED and a second dose will be given two hours prior to surgical incision.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — 2 doses of 1.95 g TXA orally, once in the ED and another dose pre-operatively.
  Arms: Tranexamic acid
Drug: Placebo — 2 doses of 1.95 g cellulose orally, once in the ED and another dose pre-operatively.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of Tranexamic acid (TXA) in reducing blood loss and transfusion requirements for patients with osteoporotic hip fractures. In addition to assessing blood loss in these patients, complications associated with TXA use would be characterized including systemic (pulmonary embolism, deep venous thrombosis, myocardial infarction, stroke) and surgical site (hematoma, infection) events, need for re-hospitalization or re-operation and 30 day mortality.

DETAILED DESCRIPTION:
Hip fractures are associated with significant blood loss and a subsequent need for blood transfusion. The causes of bleeding are multifactorial, increased fibrinolytic activity being one of them. The use of allogenic blood products is expensive and is associated with increased risk of hemolytic and anaphylactic reactions, post-operative infections and lengthened hospital stay. Tranexamic acid (TXA) is a simple and inexpensive pharmacological agent that inhibits fibrinolysis and reduced bleeding. It has a 44 year history of clinical use beginning with patients with symptomatic menorrhagia as well as bleeding prophylaxis in hemophiliac patients undergoing tooth extraction

Tranexamic acid (TXA) is an antifibrinolytic medication (reduces the destruction of blood clots, thus promoting the ability to stop bleeding) that is frequently used to reduce perioperative blood loss, blood transfusions and associated costs in major cardiac, vascular, obstetric, and orthopedic procedures. It has been used successfully in orthopedics to reduce perioperative blood loss, particularly in spine surgery, total knee and total hip arthroplasty (THA). Multiple recent meta-analyses have found that use of TXA in the setting of total knee arthroplasty (TKA) and THA leads to significantly less overall blood loss and lower rates of blood transfusion without increasing rates of venous thromboembolism (VTE) or other complications.

Osteoporotic hip fractures are at an increased risk than elective orthopaedic surgery patients because they are exposed to a double bleeding insult. Fractures bleed and many of these patients sustain their first hit when hematoma forms in their soft tissues leading to symptomatic anemia. Subsequently these patients sustain additional blood loss when they undergo surgery for definitive treatment of their injuries.

Trauma surgeons understand the risk of hemorrhage associated with trauma and routinely give TXA to patients who present with high energy injuries. The CRASH-2 trial was an international study which randomized 20,000 bleeding trauma patients to get TXA or matching placebo upon presentation. With 99.5% follow up, the authors noted a decreased risk of bleeding and death without ill effect.

However, there are limited data on its use in patients with hip fractures. We propose a double-blinded, randomized, controlled trial comparing perioperative administration of TXA to placebo in the setting of femur fractures. Thus our goal is to examine the safety and efficacy of TXA in reducing blood loss and red blood cell requirement for patients with intertrochanteric, subtrochanteric femur fractures at the time of hospital admission.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with femoral neck, intertrochanteric and subtrochanteric femur fractures Patients age 18 and older Low energy injury

Exclusion Criteria:

Pregnant or breast-feeding women Allergy to tranexamic acid Acquired disturbances of color vision Thrombophilia Antithrombin deficiency Factor V Leiden Antiphospholipid Syndrome Protein C and S deficiency History of heparin induced thrombocytopenia Sickle cell anemia Myeloproliferative disorders International Normalized Ratio (INR) > 1.4 Partial Thromboplastin Time (PTT) > 1.4 times normal A history of arterial or venous thromboembolism Cerebral Vascular Accident Deep Vein Thrombosis Pulmonary Embolism Subarachnoid hemorrhage Active intravascular clotting Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Leslie, DO, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — Study Terminated | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Loss
Time Frame: Postoperative day 3
Population: Data were not collected post surgery due to study termination.
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Hemoglobin Level
Time Frame: From presentation until postoperative day 3
Population: Data were not collected post surgery due to study termination.
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Transfusion Events
Time Frame: Postoperative day 3
Population: Data were not collected post surgery due to study termination.
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospital Length of Stay
Time Frame: During hospitalization, likely less than 1 week
Population: Data were not collected post surgery due to study termination.
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Complications
Description: Data were not collected post surgery due to study termination.
Time Frame: 6 weeks
Population: Data were not collected post surgery due to study termination.
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were not collected and analyzed due to study termination.
Description: Data, including post surgical adverse events, were not collected post surgery due to study termination.
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT02908516/Prot_SAP_000.pdf